CLINICAL TRIAL: NCT01696071
Title: A Randomised, Double- Blind, 2 Way Cross-over Study to Determine 24-hour FEV1-time Profile of Inhaled Tiotropium, Delivered Via the Respimat Inhaler, After 4 Weeks of Once Daily [5 mcg in the Evening (2 Actuations of 2.5 mcg)] or Twice Daily [2.5 mcg in the Morning and Evening (2 Actuations of 1.25 mcg)] Administration in Patients With Moderate Persistent Asthma.
Brief Title: Comparison of Two Daily Dose Regimens of Tiotropium 5 µg Once Daily and Tiotropium 2.5 µg Twice Daily for 4 Weeks on Top of Maintenance Therapy With Inhaled Corticosteroid Controller Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.441; 2012-001873-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; BID protein, human

ARMS (2):
- Treatment A (Experimental): 2 puffs of daily dose (5 mcg) in the evening and 2 puffs of matching placebo in the morning via Respimat inhaler
  Interventions: Drug: Tiotropium 5 mcg qd
- Treatment B (Experimental): 2 puffs of half daily dose (2.5 mcg) twice daily, in the evening and in the morning via Respimat inhaler
  Interventions: Drug: Tiotropium 2.5 mcg bid

INTERVENTIONS:
Drug: Tiotropium 5 mcg qd — 2 puffs (2.5 mcg each) in the evening 5 mcg in total and 2 puffs of matching placebo in the morning
  Arms: Treatment A
Drug: Tiotropium 2.5 mcg bid — 2 puffs (1.25 mcg each) twice daily, in the evening and in the morning, 5 mcg in total
  Arms: Treatment B

SUMMARY:
Determine the 24-hour FEV1-profile of tiotropium solution for inhalation after 4 weeks treatment periods of 5 mcg tiotropium administered once daily in the evening and 2.5 mcg tiotropium administered twice daily (morning and evening). In addition compare the 24 hours pharmacokinetic profile of 5 mcg tiotropium administered once daily and 2.5mcg tiotropium administered twice daily in pharmacokinetic sub-investigation.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with ICH-GCP guidelines and local legislation prior to participation in the trial.
2. Male or female patients aged at least 18 years at Visit 0 but not more than 75 years at Visit 0.
3. All patients must have at least a 3 months history of asthma at the time of enrolment (signing ICF) into the trial. The initial diagnosis of asthma must have been made before the patient's age of 40.
4. All patients must have a pre-bronchodilator FEV1 = 60% predicted and = 90% of predicted normal at Visit 1.Variation of absolute pre-bronchodilator FEV1 values at Visit 1 and Visit 2 must be within ± 30%.
5. Patient's diagnosis of asthma has to be confirmed at Visit 1 with bronchodilator reversibility (ie 10 minutes prior to and 15-30 minutes after inhalation of 400 µg salbutamol) defined as an FEV1 increase of = 12% and = 200 mL.
6. All patients must have a diagnosis of moderate persistent asthma and must be symptomatic despite their current maintenance treatment with medium doses of ICS.
7. All patients must be symptomatic at Visit 1and Visit 2 as defined by an ACQ mean score of = 1.5.
8. All patients must have maintenance treatment with stable medium daily dose of ICS for at least 4 weeks prior to Visit 1.
9. Patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment (Visit 0) and who have a smoking history of less than 10 pack-years at Visit 0.
10. Patients must be able to use the Respimat inhaler correctly.
11. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of the AM3 (e-diary) compliance of at least 80% is required.
12. Patients taking a chronic pulmonary medication allowed by the study protocol must be willing to continue this therapy for the entire duration of the study (exception: times of acute disease deterioration).

Exclusion criteria:

1. Patients with a significant disease other than asthma. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant abnormal screening hematology or blood chemistry at Visit 1 if the abnormality defines a significant disease as defined in exclusion criterion no. 1.
3. Patients requiring more than 12 puffs of rescue medication (salbutamol MDI) per 24 hours for more than 2 consecutive days between Visit 1 and Visit 2 (screening period).
4. Patients with a recent history (ie six months or less) of Acute Coronary Syndrome (STEMI, non-STEMI, Unstable Angina Pectoris) prior to Visit 1 (screening).
5. Patients who have been hospitalised for cardiac failure during the past year prior to Visit 1 (screening).
6. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year prior to Visit 1 (screening).
7. Patients with lung diseases other than asthma (eg COPD).
8. Patients with known active tuberculosis.
9. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years prior to Visit 1 (screening). Patients with treated basal cell carcinoma are allowed.
10. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no. 1.
11. Patients with significant alcohol or drug abuse on Investigator's assessment within the past two years prior to Visit 1 (screening).
12. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to Visit 1 (screening).
13. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the study medication delivery systems.
14. Pregnant or nursing women, including female patients with positive ß-HCG test at Visit 1.
15. Female patients of child-bearing potential not using highly effective method of birth control. As defined in ICH (M3) [R09-1400], note 3, highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate (ie less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner. Barrier contraceptives (eg male condom or diaphragm) are acceptable if used in combination with spermicides (eg foam, gel).

    Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation/salpingectomy, or post-menopausal for at least two years.
16. Patients who have been treated with restricted medication prior to Visit 1 and/or during the screening period.
17. Patients with any asthma exacerbation or any respiratory tract infection in the four weeks prior to Visit 1 or during the screening period.

    Visit 1 and/or Visit 2 should be postponed in case of an asthma exacerbation or respiratory tract infection. Refer to Section 6.1 for information on re-scheduling of visits.
18. Patients who are currently participating in another trial or who have been participating in another trial within one month prior to Visit 0, and patients who have previously been randomised in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (22):
- Austria (4):
  - 205.441.43004 Boehringer Ingelheim Investigational Site, Grieskirchen
  - 205.441.43003 Boehringer Ingelheim Investigational Site, Linz
  - 205.441.43001 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
  - 205.441.43002 Boehringer Ingelheim Investigational Site, Wels
- Germany (11):
  - 205.441.49015 Boehringer Ingelheim Investigational Site, Berlin
  - 205.441.49003 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.441.49014 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.441.49007 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 205.441.49005 Boehringer Ingelheim Investigational Site, Hanover
  - 205.441.49004 Boehringer Ingelheim Investigational Site, Leipzig
  - 205.441.49010 Boehringer Ingelheim Investigational Site, Lübeck
  - 205.441.49013 Boehringer Ingelheim Investigational Site, Mannheim
  - 205.441.49001 Boehringer Ingelheim Investigational Site, Neu-Isenburg
  - 205.441.49002 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 205.441.49011 Boehringer Ingelheim Investigational Site, Wiesloch
- Hungary (5):
  - 205.441.36003 Boehringer Ingelheim Investigational Site, Cegléd
  - 205.441.36002 Boehringer Ingelheim Investigational Site, Gödöllő
  - 205.441.36001 Boehringer Ingelheim Investigational Site, Pécs
  - 205.441.36005 Boehringer Ingelheim Investigational Site, Százhalombatta
  - 205.441.36004 Boehringer Ingelheim Investigational Site, Szigetszentmiklós
- Slovenia (2):
  - 205.441.38601 Boehringer Ingelheim Investigational Site, Golnik
  - 205.441.38602 Boehringer Ingelheim Investigational Site, Kamnik

RESULTS

PARTICIPANT FLOW:
Groups:
- Tio R2.5 Twice Daily (BID) / Tio R5 Once Daily (QD): Subjects were randomised to receive treatment with 2.5 μg tiotropium inhalation solution twice daily (i.e. in the morning and in the evening) and 5 μg tiotropium inhalation solution once daily in the evening via Respimat inhaler in a crossover manner using a predefined randomisation sequence.
  Treatment 1: Tio 2.5 µg BID (twice daily):Oral inhalation via the( Tiotropium-Respimat) inhaler of 2.5 µg twice daily i.e 2 actuations of 1.25 µg tiotropium in the morning and in the evening (total daily dose of 5 μg) Treatment 2: Tio 5 µg QD (once daily):Oral inhalation via the( Tiotropium-Respimat) inhaler of 5 µg once daily i.e 2 actuations of 2.5 µg tiotropium in the evening and 2 actuations of placebo in the morning (total daily dose of 5 μg)
- Tio R5 QD / Tio R2.5 BID: Subjects were randomised to receive treatment with 2.5 μg tiotropium inhalation solution twice daily (i.e. in the morning and in the evening) and 5 μg tiotropium inhalation solution once daily in the evening via Respimat inhaler in a crossover manner using a predefined randomisation sequence.
  Treatment 1: Tio 5 µg QD (once daily):Oral inhalation via the( Tiotropium-Respimat) inhaler of 5 µg once daily i.e 2 actuations of 2.5 µg tiotropium in the evening and 2 actuations of placebo in the morning (total daily dose of 5 μg) Treatment 2: Tio 2.5 µg BID (twice daily):Oral inhalation via the( Tiotropium-Respimat) inhaler of 2.5 µg twice daily i.e 2 actuations of 1.25 µg tiotropium in the morning and in the evening (total daily dose of 5 μg)
Period: Treatment Period 1: 4 Weeks
Arm/Group | Tio R2.5 Twice Daily (BID) / Tio R5 Once Daily (QD) | Tio R5 QD / Tio R2.5 BID
Started | 51 | 47
Completed | 51 | 47
Not Completed | 0 | 0
Period: Treatment Period 2: 4 Weeks
Arm/Group | Tio R2.5 Twice Daily (BID) / Tio R5 Once Daily (QD) | Tio R5 QD / Tio R2.5 BID
Started | 51 | 47
Completed | 50 | 47
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) : All patients who were dispensed study medication and were documented as having taken at least one dose of investigational treatment.
Groups:
- Baseline Total: Total number of patients randomised and treated in the study.
Arm/Group | Baseline Total
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 - 24h (AUC 0-24) Response.
Description: Mixed Model Repeated Measure (MMRM) results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres.
  The values recorded at 11 hours 50 minutes and at 23 hours 50 minutes post dosing were assigned to 12 and 24 hours, respectively.
Time Frame: Baseline FEV1 taken at visit 2 prior to the first evening dose of randomised study medication. Then, 10 minutes (min) prior to dose to 30 min,1 hour (h),2h,3h,4h,11h50min,12h30min,13h,14h,15h,16h,18h,20h,22h and 23h,23h50min relative to dose after 4 weeks
Population: Full Analysis Set (FAS): The full analysis set (FAS) includes all patients in the treated set who had baseline data and at least one on-treatment efficacy value after 4 weeks on treatment within a period.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Tio R2.5 BID: Tiotropium 2.5 mcg BID morning and evening delivered by the Respimat inhaler, on top of maintenance therapy with inhaled corticosteroid (iCS).
- Tio R5 QD: Tiotropium 5 mcg QD in the evening and matching placebo qd in the morning delivered by the Respimat inhaler, on top of maintenance therapy with iCS.
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Liters | 0.219 (0.031) | 0.217 (0.031)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.002, 95% CI [-0.038 to 0.034], Standard Error of Mean 0.018 — Tio R5 QD - Tio R2.5 BID

2. Secondary Outcome: FEV1 AUC0-12h Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC0-12h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: Baseline FEV1 taken at visit 2 prior to the first evening dose of randomised study medication. Then, 10 minutes(min) prior to dose to 30min,1hour(h),2h,3h,4h,11h50min,12h30min,13h,14h,15h,16h,18h,20h,22h and 23h,23h50min relative to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Groups:
- Tio R2.5 BID: Tiotropium 2.5 mcg BID morning and evening delivered by the Respimat inhaler, on top of maintenance therapy with iCS.
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.182 (0.031) [-0.032 to 0.052] | 0.192 (0.031) [-0.032 to 0.052]
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.010, 95% CI [-0.032 to 0.052], Standard Error of Mean 0.021 — Tio R5 qd - Tio R2.5 bid

3. Secondary Outcome: FEV1 AUC12-24h Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline. Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC12 -24h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.256 (0.033) | 0.243 (0.033)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.014, 95% CI [-0.050 to 0.022], Standard Error of Mean 0.018 — Tio R5 qd - Tio R2.5 bid

4. Secondary Outcome: Peak FEV1 Response.
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. Peak FEV1 was defined as the highest FEV1 reading observed within the 24 hour period following inhalation of the last evening dose of study medication (FEV1 Peak0-24h). The values recorded at 11 hours 50 minutes and at 23 hours 50 minutes post dosing were assigned to 12 and 24 hours, respectively.
Time Frame: 10 minutes (min) prior to dose to 30 min,1 hour (h),2h,3h,4h,11h50min,12h30min,13h,14h,15h,16h,18h,20h,22h and 23h,23h50min relative to dose after 4 weeks.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.465 (0.031) | 0.451 (0.031)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.014, 95% CI [-0.051 to 0.023], Standard Error of Mean 0.018 — Tio R5 qd - Tio R2.5 bid

5. Secondary Outcome: Trough FEV1 (L) Response.
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. Trough FEV1 was defined as the FEV1 value just prior to the last evening dose of study medication.
Time Frame: 10 minutes (min) prior to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.203 (0.033) | 0.207 (0.034)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.004, 95% CI [-0.060 to 0.068], Standard Error of Mean 0.032 — Tio R5 qd - Tio R2.5 bid

6. Secondary Outcome: Forced Vital Capacity (FVC) AUC0-24h Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres.
  The values recorded at 11 hours 50 minutes and at 23 hours 50 minutes post dosing were assigned to 12 and 24 hours, respectively.
Time Frame: Baseline taken at visit 2 prior to the first evening dose of randomised study medication. Then, 10 minutes(min) prior to dose to 30min,1hour(h),2h,3h,4h,11h50min,12h30min,13h,14h,15h,16h,18h,20h,22h and 23h,23h50min relative to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.079 (0.032) | 0.075 (0.032)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.005, 95% CI [-0.044 to 0.035], Standard Error of Mean 0.020 — Tio R5 qd - Tio R2.5 bid

7. Secondary Outcome: FVC AUC0-12h Response
Description: as for outcome 2
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.056 (0.031) | 0.053 (0.031)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.003, 95% CI [-0.048 to 0.042], Standard Error of Mean 0.023 — Tio R5 qd - Tio R2.5 bid

8. Secondary Outcome: FVC AUC12-24h Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC12 -24h calculated using the trapezoidal rule divided by the observation time (12 hours) to report in litres.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.102 (0.034) | 0.096 (0.034)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.006, 95% CI [-0.047 to 0.034], Standard Error of Mean 0.020 — Tio R5 qd - Tio R2.5 bid

9. Secondary Outcome: Peak FVC Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. Peak FVC was defined as the highest FVC reading observed within the 24 hour period following inhalation of the last evening dose of study medication (FVC Peak0-24h).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.328 (0.033) | 0.309 (0.033)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.019, 95% CI [-0.070 to 0.032], Standard Error of Mean 0.026 — Tio R5 qd - Tio R2.5 bid

10. Secondary Outcome: Trough FVC Responses
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. Trough FVC was defined as the FVC value just prior to the last evening dose of study medication.
Time Frame: Baseline taken at visit 2 prior to the first evening dose of randomised study medication. Then, 10 minutes(min) prior to dose after 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres | 0.077 (0.034) | 0.118 (0.034)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.041, 95% CI [-0.030 to 0.111], Standard Error of Mean 0.035 — Tio R5 qd - Tio R2.5 bid

11. Secondary Outcome: Peak Expiratory Flow (PEF) AUC0-24h Response
Description: MMRM results. Response was defined as change from baseline. Means are adjusted for treatment, period, patient and study baseline.Measured following the respective dosing determined at the end of each 4 week period of randomised treatment. AUC0-24h calculated using the trapezoidal rule divided by the observation time (24 hours) to report in litres per minute.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres/min
Arm/Group | Tio R2.5 BID | Tio R5 QD
Number analyzed (Participants) | 98 | 97
Litres/min | 42.788 (5.923) | 41.399 (5.933)
Statistical Analysis 1: Comparison: Tio R2.5 BID vs Tio R5 QD; No p-values are presented as no formal statistical hypothesis was tested; Test type: Superiority or Other; Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -1.389, 95% CI [-8.651 to 5.873], Standard Error of Mean 3.658 — Tio R5 qd - Tio R2.5 bid

ADVERSE EVENTS:
Time Frame: From baseline visit to end of study drug administration, plus 30 days, up to 82 days.
Arm/Group | Tio R2.5 Bid | Tio R5 qd
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/98
Other Adverse Events (participants affected / at risk) | 0/98 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tio R2.5 Bid (N=98) | Tio R5 qd (N=98)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific and statistical accuracy, within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.